CLINICAL TRIAL: NCT03828214
Title: Post Stroke Walking Kinematics Using the Honda Walking Assist Robotic Exoskeleton
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: College of St. Scholastica, Inc. (Other)
Collaborators: Honda Research and Development Americas (Industry)
Responsible Party: Principal Investigator, Alexandra Borstad, Associate Professor, College of St. Scholastica, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 001
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Stroke
Keywords: exoskeleton; gait; kinematics; EMG; stair climbing
MeSH Terms: conditions — Stroke | interventions — Exoskeleton Device

STUDY DESIGN:
Intervention Model Description: Within-subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Robotic exoskeleton for walking assist — Participants will have two testing sessions in this within-subject design experiment. The conditions under which walking will be evaluated are control (normal) walking, walking with the exoskeleton assistance and walking immediately following exoskeleton walking. The conditions under which stair walking (ascending and descending) will be evaluated include control (normal) stairs and exoskeleton assisted stairs. Assistance is provided by The Honda Walking Assist (HWA) System is a robotic device developed by Honda R&D Corporation ®, Japan. The devices computer-activated motors use hip angle information to guide assistance delivered through the thigh straps to the legs in time with the walking cycle. The maximum torque delivered is 4 Newton-meters.

SUMMARY:
To investigate the effect of a robotic exoskeleton on kinematics, muscle activity, ground reaction forces and spatiotemporal characteristics during walking in persons post stroke.

DETAILED DESCRIPTION:
Following stroke walking dysfunction is prevalent. Traditional rehabilitation methods fall short of achieving desirable walking outcomes for most people who experience stroke. Robotic methods to assist walking, such as the Honda Walking Assist Device (HWA) Robot from Honda R & D Americas Inc., are being explored as a means of improving the recovery of walking post stroke. Prior to examining the effectiveness of exoskeletal robots for walking recovery it is important to understand their effect on kinematic and muscle responses during walking. Kinematic and muscle responses at the hip during walking with the HWA were recently described.

The purpose of this study is to quantify the effect of walking with the HWA on body segments remote from the hip. These segments include knee, ankle, trunk and arm. The non-invasive measures used will include: walking kinematics (measurement of joint angles using cameras), muscle activity (Electromyography), ground reaction forces (detected by a force plate in the floor) and spatiotemporal characteristics (such as walking speed). Measures will be collected under three conditions: 1) walking at self-selected pace (control), 2) walking at self-selected pace with the HWA (4 Newton-meter assist mode for hip flexion and extension), 3) walking immediately following HWA use (aftereffect).

ELIGIBILITY:
Inclusion Criteria:

* ≥12 weeks but <1 year post stroke at time of study participation
* Age: 18-85 years
* Ability to walk a minimum of 10 meters with standby assistance with or without orthosis or assistive device (Functional Ambulation categories 3, 4 or 5)
* Able to follow three step commands
* Express the ability to understand study tasks and purpose
* Able and willing to provide written informed consent
* Living in the community with the ability to travel to maurices Community Clinic for testing
* Willingness to wear the StepWatch pedometer for a period of 3 days in their home
* (If applicable) ≥ 90 days post major orthopedic surgery (such as a joint replacement)
* (If applicable) ≥ 6 months post cardiac surgery

Exclusion Criteria:

* Serious cardiac conditions (hospitalized for myocardial infarction or heart surgery within 3 months, congestive heart failure, unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living)
* Severe arthritis or orthopedic conditions that limit lower extremity range of motion (> 10° or < 90° knee flexion, lacking > 25° hip extension, >15° from neutral plantar flexion.)
* Preexisting neurologic disorders such as Dementia, Multiple Sclerosis, Amyotrophic Lateral Sclerosis, Parkinson's Disease or Ataxia.
* History of lower limb amputation, non-healing ulcers, legal blindness or severe visual impairment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra L Borstad, PhD, Principal Investigator — College of St. Scholastica
Locations (1):
- College of St. Scholastica-Health Science Center, Duluth, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Walking: In this study a single group of participants were observed in each of 4 conditions: control walking (CI), HWA walking (C2), Aftereffect (C3), and Late aftereffect (C4)
Period: Overall Study
Arm/Group | Walking
Started | 11
Completed | 11 (11 participants completed this study, however, for some outcome variables, only data from 9 or 10 participants was available for analysis due to technical challenges during data collection.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Walking: In this study a single group of participants were studied during one session in each of 4 conditions: control walking (CI), HWA walking (C2), Aftereffect (C3), and Late aftereffect (C4)
Arm/Group | Walking
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Height [Mean (Standard Deviation); unit: cm] | 163 (9.4)
weight [Mean (Standard Deviation); unit: kg] | 81 (22.2)
Stroke affected side was left [Count of Participants; unit: Participants] | 9
Time post stroke [Mean (Standard Deviation); unit: months] | 7.3 (4)
Fugl-meyer Assessment [Mean (Standard Deviation); unit: units on a scale] — The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index.
  For this study the FM Lower extremity subset was used to characterize participants. Scores on this subset could range from 0-34 points. Higher scores indicate less lower extremity impairment.
  units on a scale | 30.5 (1.5)
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is a cognitive screening test designed to assist Health Professionals in the detection of mild cognitive impairment and Alzheimer's disease. The total possible score is 30 points. Greater than or equal to 26 is considered normal cognitive function for an adult.
  units on a scale | 22.4 (4.3)
Activities Specific Balance Confidence Scale [Mean (Standard Deviation); unit: units on a scale] — The ABC Scale is a 16 item self-report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness. For each item participants rate them selves from 0 (no confidence) to 100 (complete confidence). The total score is an average across the 16 items.
  units on a scale | 72.9 (20.2)
Steps per day [Mean (Standard Deviation); unit: steps] — Average steps from a 3 day sample quantified using StepWatch.
  steps | 2783 (1512)

OUTCOME MEASURES:

1. Primary Outcome: Gait Kinematics
Description: Difference in affected leg maximum knee flexion angle (initial swing to midswing) between conditions Kinematic Analysis of Gait will be obtained using a Qualisys 8-camera motion capture system. Sample rate 120 Hz. A modified Istituti Ortopedici Rizzoli (IOR) gait marker set (~40 markers) applied bilaterally.
Time Frame: Gait kinematics were measured in each of 4 conditions during one 2-hour session for each participant.
Population: For one participant data was not available for the C3 condition
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Walking
Number analyzed (Participants) | 10
degrees
  C1 | 55.9 (12.3)
  C2 | 57.8 (12.4)
  C3: number analyzed (Participants) | 9
  C3 | 58.3 (8.1)
  C4 | 56.6 (12.6)
Statistical Analysis 1: Comparison: Walking; C2, C3, C4 were compared to C1 the comparison condition; Test type: Superiority; p = 0.973, ANOVA — a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 2.4, Standard Deviation 9.2

2. Secondary Outcome: Lower Limb Electromyography (EMG)
Description: Average max EMG of affected tibialis anterior muscle measured during swing phase for walking conditions using Delsys Tringo EMG sensors. Sample rate 2000Hz.
Time Frame: Measured during swing phase of gait during each of 4 walking conditions during a single data collection session.
Population: There was a single group that participated in this within subject design study, here we compare the outcome parameter across the four conditions for this group.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Walking
Number analyzed (Participants) | 10
mV
  C1 | 0.115 (0.080)
  C2 | 0.115 (0.077)
  C3 | 0.101 (0.064)
  C4 | 0.119 (0.077)

3. Secondary Outcome: Ground Reaction Force at Terminal Stance
Description: 2 Force platforms were used to quantify ground reaction forces at terminal stance for the affected lower limbs during gait. Sample rate 1200Hz.
Time Frame: Force data will be measured at a single time point (in one 2-hour session) for each participant in each of 4 conditions.
Population: n=9 for grf data 1 participant No HWA condition secondary to device slipping, 1 participant no clean force plate hits due to short step length.
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | Walking
Number analyzed (Participants) | 9
percentage of body weight
  C1 | 103 (16)
  C2 | 105 (9)
  C3 | 104 (9)
  C4 | 105 (10)

4. Secondary Outcome: Stair Climbing Ascend/Descend Test
Description: A timed test of the ability to ascend and descend stairs with our without a rail. For this study a flight of 7 stairs will be used. The means of two trials of ascending and descending will be recorded. (Flansbjer et al., 2005)
Time Frame: Stairs will be measured at a single time point (in one 2-hour session) for each participant
Measure: Mean (Inter-Quartile Range); unit: seconds
Arm/Group | Walking
Number analyzed (Participants) | 11
seconds
  ascend (control) | 7.03 [4.2 to 11]
  decend (control) | 7.61 [4 to 10.5]
  ascend with HWA | 7.10 [4 to 11]
  descend with HWA | 7.99 [4.1 to 9.5]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the one day period of participation in the study.
Arm/Group | Walking
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT03828214/Prot_SAP_000.pdf